CLINICAL TRIAL: NCT06539299
Title: Socket Preservation - How Successful is the Method for Inexperienced Practitioners? A Randomized Clinical Implementation in a Student Setting
Brief Title: Socket Preservation - A Randomized Clinical Implementation in a Student Setting
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sigmund Freud PrivatUniversitat (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SocketPreservationStudents
Record Dates: First submitted 2024-08-01; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Alveolar Bone Loss; Dental Implant; Bone Augmentation
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): No bone preservation procedure after tooth extraction
- Socket Preservation - Student (Active Comparator): Socket preservation done by a student
  Interventions: Procedure: Socket Preservation
- Socket Preservation - surgeon (Active Comparator): Socket preservation done by a surgeon
  Interventions: Procedure: Socket Preservation

INTERVENTIONS:
Procedure: Socket Preservation — After extracting a tooth, the alveolar socket is cleaned. A bone replacement material (Bio-Oss Collagen) is then placed into the socket and sutured with a collagen membrane (Mucograft-Seal). Patients will receive Antibiotics (Augmentin 875mg/125mg OR Dalacin C 300mg) and pain medication (Seractil forte 400 mg). Patients will be advised to carefully rinse with Chlorhexamed forte for one week. Sutures will be removed after two weeks.
  Arms: Socket Preservation - Student; Socket Preservation - surgeon

SUMMARY:
Preserving the ridge dimension after tooth extraction aims to avoid the need for bone augmentation procedures before implant placement. This study aims to show that socket preservation procedure is a safe, easy and predictable method that stabilizes the bone situation when late implantation is planned.

DETAILED DESCRIPTION:
Preserving the ridge dimension after tooth extraction aims to avoid the need for further augmentative procedures before implant placement. Immediately after the extraction a bone replacement material is inserted into the empty socket and covered with a membrane to protect it to maintain or even improve alveolar bone dimension. But how promising is it, if such an operation is carried out by an inexperienced practitioner? The aim is to show that socket preservation is a predictable, promising and an easy-to-implement method that creates a better initial bone situation for later implant placement. The execution by a student is intended as a simulation of a inexperienced practitioners.

Design:

A total of 51 patients with the need of extraction of a single-rooted lower jaw tooth (35-45) will be recruited from the dental clinic of the Sigmund Freud Private University. Written consent will be given before enrollment in the study. All subjects will receive a professional cleaning and hygiene instruction before the start of the study. The extracted tooth will be replaced by a dental implant after six months of healing.

The patients are divided into three groups (17 participants each).

Group 1 serves as a control group, no ridge prophylactic measures are taken after tooth extraction.

In groups 2 and 3 after the extraction, a socket preservation is made with a company's bone replacement material and a membrane (Geistlich (BioOss Collagen + Mucograft Seal)) by a student (Group 2) or investigator doctor (3. The allocation to the respective group is carried out randomly using a random generator. The entire treatment takes place in all groups under the supervision of one study doctor.

Dimensional changes of the bone will be measured after the extraction and after 6 month using CBCT Scans.

ELIGIBILITY:
Inclusion Criteria:

* Study participants have signed patient information and consent form
* Age between 18-65 years, all genders included
* Study participants who are considering a planned extraction of a mandibular posterior tooth with subsequent treatment with an implant
* Study participants with medical and anatomical conditions that correspond to the applicable instructions for use
* Study participants agree to student treatment

Exclusion Criteria:

* Study participants under 18 years of age
* Study participants with allergies or undesirable reactions to the materials used - Patients with uncontrolled diabetes mellitus (HbA1C value >8%)
* Heavy smokers (>10 cigs/day)
* Previous general medical conditions that influence bone metabolism (Bone metabolic diseases such as osteopetrosis, osteomalacia, Paget's disease, metabolic diseases such as hyperthyroidism, renal osteopathy, oophorectomy, uncontrolled diabetes mellitus type 2), malignant neoplasms, chemotherapy/radiation therapy in the head and neck area and immunocompromised patients)
* which can be determined clinically or radiologically pathological symptoms in the oral cavity or on the alveolar processes or the adjacent regions, untreated acute or chronic disease of the periodontium, untreated disease of the oral mucosa - drug abuse, alcohol disease or abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
three-dimensional bone changes | measured after six months after extraction
  horizontal bone dimension changes
three-dimensional bone changes | measured after six months
  vertical bone dimension changes

IPD SHARING:
Plan to Share IPD: No